CLINICAL TRIAL: NCT05835167
Title: Minimally Invasive Coronary Artery Bypass Grafting Achieving Complete Revascularization of Multivessel Coronary Artery Disease Via Inferior Part-Sternotomy (The ACRIS-MICABG Trial)
Brief Title: Complete Revascularization Via Inferior Part-sternotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Tangshan Central Hospital (Other); Baotou Central Hospital (Other); Xiamen Second Hospital (Unknown); Beijing Shijitan Hospital, Capital Medical University (Other); Peking University International Hospital (Other); Shenzhen Sun Yat-sen Cardiovascular Hospital (Other); Fuwai Yunnan Cardiovascular Hospital (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-GSP-GG-23
Record Dates: First submitted 2023-04-16; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Complete Revascularization; Coronary Artery Bypass Grafting; Multivessel Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inferior part-sternotomy CABG (Experimental): A midline skin incision of 8 to 10cm in length is made over the sternum, starting from 2-3cm below the sternal angle inferiorly and extending slightly beyond the xiphoid process. A sternal saw is used to split the sternum from the xiphoid process to the second intercostal space where the sternum is partially transected by turning the saw rightward. Left internal mammary artery (LIMA)-left anterior descending branch bypass is the first choice for all patients. Remaining coronary bypassing techniques are according to clinical practice and preference of the operator. If it is difficult to perform CABG via inferior part-sternotomy, the treatment strategy convert to full median sternotomy, which is deemed to be failed to achieve complete revascularization via inferior part-sternotomy.
  Interventions: Procedure: Inferior part-sternotomy
- Full median sternotomy CABG (Active Comparator): A midline skin incision is made over the sternum, starting from the sternal angle and extending slightly beyond the xiphoid process. The sternum is fully split by a sternal saw. Remaining coronary bypassing techniques are same in both groups according to clinical practice and preference of the operator.
  Interventions: Procedure: Full median sternotomy

INTERVENTIONS:
Procedure: Inferior part-sternotomy — A midline skin incision of 8 to 10cm in length is made over the sternum, starting from 2-3cm below the sternal angle inferiorly and extending slightly beyond the xiphoid process. A sternal saw is used to split the sternum from the xiphoid process to the second intercostal space where the sternum is partially transected by turning the saw rightward.
  Arms: Inferior part-sternotomy CABG
Procedure: Full median sternotomy — A midline skin incision is made over the sternum, starting from the sternal angle and extending slightly beyond the xiphoid process. The sternum is fully split by a sternal saw.
  Arms: Full median sternotomy CABG

SUMMARY:
To verify the effectiveness and safety of minimally invasive coronary artery bypass grafting for complete revascularization of multivessel coronary artery disease via inferior part-sternotomy, We aim to randomize 260 patients undergoing isolated Coronary artery bypass grafting (CABG) to compare the ratios of complete revascularization between inferior part-sternotomy CABG and full median sternotomy CABG from 9 hospitals in China.

DETAILED DESCRIPTION:
Coronary artery bypass grafting (CABG) has always been the gold standard for surgical treatment of coronary artery disease (CAD), especially for left main (LM) coronary disease, patients with high SYNTAX scores, and diabetes mellitus. By minimally invasive strategy, patients recover significantly faster in the early post-operative period. However, a prospective randomized controlled trials is needed to compare the ratios of complete revascularization between inferior part-sternotomy CABG and full median sternotomy CABG.

Objectives:

To verify the effectiveness and safety of minimally invasive coronary artery bypass grafting for complete revascularization of multivessel coronary artery disease via inferior part-sternotomy.

Study design:

This is a prospective, multicenter, open-label, randomized controlled trial. We aim to randomize 260 patients undergoing isolated CABG to compare the ratios of complete revascularization between inferior part-sternotomy CABG and full median sternotomy CABG from 9 hospitals in China. We consecutively screen patients during the study enrollment period and seek informed consent from all eligible patients. Patients who give informed consent are randomly assigned to undergo inferior part-sternotomy CABG or full median sternotomy CABG by a central randomization system. An expert group composed of three doctors with CABG qualifications will develop a plan achieving complete revascularization by coronary angiography images before the operation, including the number and location of proximal and distal anastomoses. The actual bypass procedure will be recorded and compared with the preoperative plan. We will follow-up participants until 10 years after the operation. To reduce the variation among surgeons, we require that all CABG are performed by qualified surgeons. The surgeons in this study needs to have experience in at least 100 cases of full median sternotomy CABG, and at least 5 cases of inferior part-sternotomy CABG.The ethics committees at all 9 participating hospitals approved this study.

Randomization A web-based central randomization system incorporated in the registration system is used for allocation (http://ccsr.cvs-china.com/). The randomization code with fixed block size is generated by SAS. Randomization is stratified by investigation center. When an eligible patient gives informed consent, the investigator logs in to the randomization webpage and obtain the random number along with treatment group (Inferior part-sternotomy or Full median sternotomy group) automatically distributed by the system after the basic patient information be confirmed. The statistician responsible for the randomization code and the staff who develops the Interactive Web-based Response (IWR) system are independent of each other.

Intervention Surgical procedure.The patient is placed in the supine position. Standard intubation and hemodynamic monitoring are used. Heparinization is standardized for on-pump CABG. The surgeon is given discretion to ensure that his choice in surgery would ensure the patient´s safety (including which graft to use or the choice of anatomic regions to revascularize). The surgeries are performed with the usual methods of cardiopulmonary bypass (CPB) with aortic cross-clamp technique. Myocardial protection strategies include blood cardioplegia and moderate hypothermia. For both types of surgeries, an excellent exposure is required.

Inferior part-sternotomy CABG.A sternal saw is used to split the sternum from the xiphoid process to the second intercostal space where the sternum is partially transected by turning the saw rightward. Remaining coronary bypassing techniques are same in both groups according to clinical practice and preference of the operator.

Full median sternotomy CABG. A midline skin incision is made over the sternum, starting from the sternal angle and extending slightly beyond the xiphoid process. The sternum is fully split by a sternal saw.

Medication. All participants are prescribed dual antiplatelet therapy with aspirin 100 mg plus clopidogrel 75 mg daily from the first day post-CABG until 3 months post-operation. Prescription of other concomitant medications such as β-blockers, statins, and antihypertensive agents is determined by local surgeons according to ACC/AHA guidelines.

The trial data will be analyzed on an intention-to-treat basis with patients included in the groups assigned at randomization, irrespective of future management and events.Demographic and clinical variables will be summarized as means (SDs) for continuous and counts (percentages) for categorical variables. Comparisons across the groups will be performed using a 2-tailed unpaired t test for continuous variables and the Pearson's χ2 test for categorical variables. A P value of less than 0.05 will be considered as statistically significant for all analyses.

Clinical events committee. All clinical events including myocardial infarction, stroke, target lesion revascularization, and death will undergo central adjudication by an independent clinical events committee (CEC).

ELIGIBILITY:
Inclusion Criteria:

Patients who undergo primary isolated open-chest CABG with multi-vessel coronary disease(left main artery disease with right coronary artery disease,or three-vessel disease)

Exclusion Criteria:

1. Single vessel disease, double vessel disease, left main artery disease without right coronary artery disease.
2. Concomitant cardiac surgeries(i.e. valve repair or replacement, Maze surgery, left ventricular repair due to ventricular aneurysm).
3. Redo CABG.
4. Emergent CABG.
5. Left ventricular ejection fraction(EF≤35%).
6. Severe atherosclerosis of the ascending aorta.
7. Subjects tend to choose surgical approach (via full median sternotomy/inferior part-sternotomy) .
8. Malignant tumor or other severe systemic diseases.
9. Severe renal insufficiency (i.e. creatinine >200 μmol/L).
10. Contraindications for dual antiplatelet therapy, such as active gastroduodenal ulcer.
11. Participant of other ongoing clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-05-05 (Estimated); Primary Completion 2025-05-04 (Estimated); Study Completion 2035-05-04 (Estimated)

PRIMARY OUTCOMES:
Complete revascularization rate immediately after surgery | Immediately after surgery
  Most surgical groups have adopted the functional definition in their studies. We therefore elected to use a functional definition for complete revascularization in the present study. The coronary vascular tree was divided into 3 separate territories: the left anterior descending artery (LAD), the circumflex artery, and the right coronary artery (RCA).Functional completeness of revascularization is defined as all viable myocardial territories are reperfused, as at least one bypass graft for every diseased primary arterial territory

SECONDARY OUTCOMES:
The harvest time of left Internal mammary artery (LIMA) | During surgery
  It is defined as the time from skin incision to clamping of the distal part of the LIMA.
Aortic cross-clamp time | During surgery
Overall operation time | During surgery
  It is defined as the time from skin incision to skin sutured.
Intraoperative real-time blood flow at each anastomosis | During surgery
  It was evaluated intraoperatively using ultrasound flow measurements.
The total amount of postoperative chest tube drainage | Up to 4 weeks
  This includes the amount of fluid of closed thoracic drainage or thoracentesis drainage due to pleural effusion during hospitalization.
The graft patency rate by CTA at 5-7 days, 1 year, 3 years, 5 years, and 10 years after surgery | 1week after the surgery；10 years after surgery
  Graft occlusion is detected by computed tomography angiography (CTA). Grafts are graded into three levels: A (excellent), B (fair), or C (occluded). Contrast filling of the grafts, anastomoses, and coronary arteries beyond the graft are considered in each assessment. Grade A indicates that the graft is patent with ≤50% stenosis. Grade B indicates that graft stenosis is >50% but not occluded. When a graft does not fill with contrast at all, it is considered Grade C and included with string sign found in any segment (including proximal and distal anastomotic site, and main trunk). Both of these findings are considered together and referred to as occlusion in the analysis.The patency rate of grafts = number of grafts in grades A and B/total number of bypass grafts.
The rate of major adverse cardiac or cerebrovascular events (MACCE) at 5-7 days, 1 year, 3 years, 5 years, and 10 years after surgery | 1week after the surgery；10 years after surgery
  MACCE: cardiac death, myocardial infarction, stroke, repeat revascularization and hospitalization for heart failure.
  Myocardial infarction (troponin values >10 times the 99th percentile of upper reference limit in association with new Q waves).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Lapierre H, Chan V, Sohmer B, Mesana TG, Ruel M. Minimally invasive coronary artery bypass grafting via a small thoracotomy versus off-pump: a case-matched study. Eur J Cardiothorac Surg. 2011 Oct;40(4):804-10. doi: 10.1016/j.ejcts.2011.01.066. Epub 2011 Mar 9. PMID 21393011
- [Background] Ong AT, Serruys PW. Complete revascularization: coronary artery bypass graft surgery versus percutaneous coronary intervention. Circulation. 2006 Jul 18;114(3):249-55. doi: 10.1161/CIRCULATIONAHA.106.614420. No abstract available. PMID 16847164
- [Background] Veiga Oliveira P, Madeira M, Ranchordas S, Marques M, Almeida M, Sousa-Uva M, Abecasis M, Neves JP. Complete surgical revascularization: Different definitions, same impact? J Card Surg. 2021 Dec;36(12):4497-4502. doi: 10.1111/jocs.15986. Epub 2021 Sep 16. PMID 34533240
- [Background] Sohn SH, Kang Y, Kim JS, Paeng JC, Hwang HY. Impact of Functional vs Anatomic Complete Revascularization in Coronary Artery Bypass Grafting. Ann Thorac Surg. 2023 Apr;115(4):905-912. doi: 10.1016/j.athoracsur.2022.10.029. Epub 2022 Nov 9. PMID 36334649
- [Background] Sun HS, Ma WG, Xu JP, Sun LZ, Lu F, Zhu XD. Minimal access heart surgery via lower ministernotomy: experience in 460 cases. Asian Cardiovasc Thorac Ann. 2006 Apr;14(2):109-13. doi: 10.1177/021849230601400206. PMID 16551816
- [Background] Kleisli T, Cheng W, Jacobs MJ, Mirocha J, Derobertis MA, Kass RM, Blanche C, Fontana GP, Raissi SS, Magliato KE, Trento A. In the current era, complete revascularization improves survival after coronary artery bypass surgery. J Thorac Cardiovasc Surg. 2005 Jun;129(6):1283-91. doi: 10.1016/j.jtcvs.2004.12.034. PMID 15942568